CLINICAL TRIAL: NCT05729685
Title: Aerobic Adaptations Following Two Iso-effort Training Programs: An Intense Continuous and a High-intensity Interval
Brief Title: Aerobic Adaptations With Various Training Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ilias Smilios (Other)
Responsible Party: Sponsor-Investigator, Ilias Smilios, Associate Professor, Democritus University of Thrace
Organization: Democritus University of Thrace (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AERCONINT
Record Dates: First submitted 2023-01-26; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: exercise; maximal oxygen consumption; endurance
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: A parallel group research design was used in the present study. Initially, 26 participants (10 males and 16 females), using stratified randomization (gender was the variable of stratification) were randomly assigned (1:1), according to a random-number table, either to an intense continuous training group (CON) or to a high-intensity interval training group (INT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interval training (Experimental): The interval group trained using the interval trainining method.
  Interventions: Other: Interval training
- Continuous training (Experimental): The continuous group trained using the continuous training method.
  Interventions: Other: Continuous training

INTERVENTIONS:
Other: Interval training — The interval training group trained using the interval method. During the exercise sessions the participants ran each bout at an intensity corresponding to 90% of PTV. PTV was used to prescribe the exercise intensity at the INT group. The duration of the running-bouts was equal to ¼ of the individual time to exhaustion at 90% of PTV (determined during the CV testing) followed by passive rest equal to 2/3 of exercise duration. The duration of the exercise-bouts was individualized based on the time to exhaustion at 90% of PTV to reduce the between subject's variability. The participants terminated each exercise session when an RPE value of 17 was reached. Running bout duration and intensity were adjusted after 7 training sessions (during the 3rd week) following a reassessment of the time to exhaustion at 90% of the "new" PTV achieved during mid-testing as a result of training.
  Arms: Interval training
Other: Continuous training — The continuous group trained using the continuous method. During the training sessions the participants ran with an intensity corresponding to -2,5% of CV until they reported a rating of 17 at the 6-20 Borg's scale. Running velocity was adjusted after 7 training sessions (during the 3rd week) after reassessment of CV. CV was used to determine the exercise intensity in the CONT group to ensure that all individuals would ran at the heavy intensity domain and be able to complete at least 15 min of continuous running, and to minimize the high inter-individual variations in endurance time at intensities near the upper limit of the heavy intensity domain. Using PTV to determine the intensity in the CONT group, would increase the possibility for trainees to exercise at different exercise intensity domains.
  Arms: Continuous training

SUMMARY:
The goal of this intervention study is to compare the adaptations after a 6-week training period between an intense continuous and a high-intensity interval training program performed under iso-effort conditions on aerobic performance parameters in young healthy adults. The main question it aims to answer are if the intense continuous and a high-intensity interval training programs will induce similar adaptations in maximal (VO2max and PTV) and submaximal (critical velocity, lactate threshold parameters and running economy) aerobic performance parameters. Participants will be ere randomly assigned either to an intense continuous training group (CON) or to a high-intensity interval training group (INT). The training program will comprise of 14 training sessions performed over a 6-week period.

DETAILED DESCRIPTION:
The aim of this study was to compare the adaptations after a 6-week training period between the intense continuous and the high-intensity interval training methods performed under iso-effort conditions on maximal (VO2max and PTV) and submaximal (critical velocity, lactate threshold parameters and running economy) aerobic performance parameters.

A parallel group research design was used in the present study. Initially, 26 participants (10 males and 16 females), using stratified randomization (gender was the variable of stratification) were randomly assigned (1:1), according to a random-number table, either to an intense continuous training group (CON) or to a high-intensity interval training group (INT).

The INT group trained using the interval method. During the exercise sessions the participants ran each bout at an intensity corresponding to 90% of PTV. PTV was used to prescribe the exercise intensity at the INT group. The duration of the running-bouts was equal to ¼ of the individual time to exhaustion at 90% of PTV (determined during the CV testing) followed by passive rest equal to 2/3 of exercise duration. The duration of the exercise-bouts was individualized based on the time to exhaustion at 90% of PTV to reduce the between subject's variability. The participants terminated each exercise session when an RPE value of 17 was reached. Running bout duration and intensity were adjusted after 7 training sessions (during the 3rd week) following a reassessment of the time to exhaustion at 90% of the "new" PTV achieved during mid-testing as a result of training.

The CONT group trained using the continuous method. During the training sessions the participants ran with an intensity corresponding to -2,5% of CV until they reported a rating of 17 at the 6-20 Borg's scale. Running velocity was adjusted after 7 training sessions (during the 3rd week) after reassessment of CV. CV was used to determine the exercise intensity in the CONT group to ensure that all individuals would ran at the heavy intensity domain and be able to complete at least 15 min of continuous running, and to minimize the high inter-individual variations in endurance time at intensities near the upper limit of the heavy intensity domain. Using PTV to determine the intensity in the CONT group, would increase the possibility for trainees to exercise at different exercise intensity domains.

During the experiment, participants will not perform any other form of training besides of that applied in the current study. VO2max, PTV, oxygen consumptions, heart rates and the velocities corresponding to the 1st and the 2nd lactate thresholds (LT1 and LT2), the velocity at 4 mmol/L of blood lactate concentration (v4mmol), running economy, and critical velocity (CV) will be measured before, after 7 training sessions (3rd week, two days after the 7th training session), and after the completion of training program.

ELIGIBILITY:
Inclusion criteria

* All participants should have been involved in low intensity continuous training,
* All participants should have been training 1-3 times per week for 30-45 min for at least three months.

Exclusion criteria

* Not familiar with aerobic training
* Any health issues that did not allow participation in regular exercise training.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Changes in maximal oxygen consumption | At the beginning of the training program, the 3rd week of training (after 7 training sessions), and the 7th week after the start of the intervention (after the completion of 6 weeks of training, 14 training sessions)
  Maximal oxygen consumption in ml/kg/min
Changes in peak treadmill velocity | At the beginning of the training program, the 3rd week of training (after 7 training sessions), and the 7th week after the start of the intervention (after the completion of 6 weeks of training, 14 training sessions)
  Peak treadmill velocity using a maximal incremental test to exhaustion on a treadmill in km/h
Changes in running velocities at the 1st and the 2nd lactate thresholds | At the beginning of the training program, the 3rd week of training (after 7 training sessions), and the 7th week after the start of the intervention (after the completion of 6 weeks of training, 14 training sessions)
  Running velocities (km/h) at the 1st and the 2nd lactate thresholds by measuring the changes in blood lactate concentration during a maximal incremental test to exhaustion on a treadmill.
Changes in critical velocity | At the beginning of the training program, the 3rd week of training (after 7 training sessions), and the 7th week after the start of the intervention (after the completion of 6 weeks of training, 14 training sessions)
  Critical velocity (km/h) determined by having the participants ran until exhaustion at velocities corresponding to 90, 100, and 110% of peak treadmill velocity. Using linear regression analyses, the relationship between the distance covered at each run and the time to exhaustion was calculated. Τhe slope of the linear regression line was the critical velocity.

SECONDARY OUTCOMES:
Changes in running economy | At the beginning of the training program and the 7th week after the start of the intervention (after the completion of 6 weeks of training, 14 training sessions)
  Running economy determined by measuring the oxygen consumption (ml/kg/min) while running for 10 min at a velocity corresponding to 70% of the pre-training peak treadmill velocity
Changes in running velocity at a blood lactate concentration of 4 mmol/L | At the beginning of the training program and the 7th week after the start of the intervention (after the completion of 6 weeks of training, 14 training sessions)
  Running velocity (km/h) at a blood lactate concentration of 4 mmol/L determined by the individual relationship between lactate concentrations and running velocities during an incremental test by applying a nonlinear regression model.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Education and Sport Science, Komotini, Rodopi, Greece

IPD SHARING:
Plan to Share IPD: No